CLINICAL TRIAL: NCT06489015
Title: An Open-label, Parallel-group Exploratory Clinical Trial to Evaluate the Safety and Preliminary Efficacy of Recombinant Human Serum Albumin Injection in the Treatment of Mild to Moderate Alzheimer's Disease
Brief Title: Recombinant Human Serum Albumin in the Treatment of AD (Alzheimer Disease) Exploratory Clinical Trials
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Protgen Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rHSA2024-01
Record Dates: First submitted 2024-06-26; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer's Disease (AD)
MeSH Terms: conditions — Alzheimer Disease | interventions — recombinant human serum albumin-heme

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 20g dose group (Experimental)
  Interventions: Drug: Recombinant Human Serum Albumin
- 30g dose group (Experimental)
  Interventions: Drug: Recombinant Human Serum Albumin
- 40g dose group (Experimental)
  Interventions: Drug: Recombinant Human Serum Albumin

INTERVENTIONS:
Drug: Recombinant Human Serum Albumin — Each group receives the investigational drug (recombinant human serum albumin), with the distinction being the variation in dosing.

SUMMARY:
This clinical trial is an open-label, parallel-group, exploratory study of recombinant human serum albumin (rHSA, hereafter referred to as the "investigational drug") in patients with mild to moderate Alzheimer's Disease (AD). It aims to enroll 30 subjects who meet the 2011 National Institute on Aging and Alzheimer's Association (NIA-AA) criteria for "Probable AD Dementia." Participants will be randomized in a 1:1:1 ratio to receive the investigational drug at doses of 20g, 30g, or 40g, for assessments of safety and preliminary efficacy. Stratification factors will be based on the severity classification (mild; moderate) as indicated by the total score on the Clinical Dementia Rating Scale - Global Score (CDR-GS) during the screening period.

ELIGIBILITY:
Inclusion Criteria：

1. Aged between 50 and 85 years (inclusive), with no gender restrictions;
2. Meet the 2011 National Institute on Aging and Alzheimer's Association (NIA-AA) criteria for "Probable AD Dementia";
3. Mild to moderate disease stage, as indicated by a Clinical Dementia Rating Scale - Global Score (CDR-GS) ≤ 2;
4. Hachinski Ischemia Scale (HIS) ≤ 4;
5. Geriatric Depression Scale (GDS) score between 0 and 10 (inclusive);
6. Memory impairment present for at least 12 months with evidence of progression;
7. Availability of a qualified brain MRI scan within 1 month prior to enrollment, or willingness to undergo an MRI scan, showing: No more than 2 infarcts larger than 2 cm, no infarcts in key areas such as the thalamus, hippocampus, entorhinal cortex, perirhinal cortex, angular gyrus, cortical or subcortical gray matter nuclei, and imaging features highly suggestive of Alzheimer's Disease (Medial Temporal Lobe Atrophy [MTA] scale rating ≥ 2);
8. Female participants must be postmenopausal for at least 24 weeks, have undergone sterilization surgery, or if of childbearing potential, along with fertile males, agree to use effective contraception during the study. Women of childbearing potential or those postmenopausal for less than 24 weeks require a negative pregnancy test at screening;
9. If patients were on Alzheimer's medications such as cholinesterase inhibitors, NMDA receptor antagonists, or Oligomannate capsules, or taking other drugs that could affect cognition (e.g., Ginkgo biloba, Ginkgo leaf extract, Vitamin E, Selegiline, Folic acid, Estrogen, traditional Chinese medicines including compound sea snake capsules, Citicoline, Piracetam, Aniracetam, etc.), they must have been on a stable dose for at least 30 days before screening, with the investigator determining suitability and the patient agreeing to maintain this stable dose throughout the trial;
10. Patients must have a stable and dependable caregiver or adequate care arrangements (a minimum of 4 days weekly, 2 hours daily), with the caregiver willing to assist in the patient's full participation in the trial, including accompanying them to visits and helping with assessment scales;
11. Patients should have an educational level of primary school completion or above, capable of completing cognitive assessments and other tests as required by the protocol;
12. Written informed consent obtained.

Exclusion Criteria:

1. Dementia secondary to other causes: frontotemporal dementia, dementia with Lewy bodies, vascular dementia, Parkinson's disease dementia, dementia due to epilepsy, post-traumatic dementia, central nervous system infections, and immune-mediated dementias, among others;
2. Known history of allergy or allergic reactions to yeast or yeast-derived products, any component of the study formulation, individuals with an allergic constitution (multiple drug or food allergies), a history of severe systemic allergic reactions to biologics, or those deemed unsuitable for trial drug treatment by the investigator;
3. Active or historical cardiovascular disorders at screening or conditions deemed inappropriate for human albumin treatment by the investigator, specifically including but not limited to: hypertension (systolic blood pressure >160 mmHg or diastolic >100 mmHg, unless well-controlled with medication and stable in the investigator's judgment), severe anemia, acute cardiac events, significant heart or pulmonary structural diseases, severe arrhythmias, decompensated heart failure (in normal or high volume states), unstable angina, myocardial infarction within 6 months prior to screening, medically treated tachycardia/bradycardia, third-degree atrioventricular block, etc.;
4. Active metabolic disorders or history thereof at screening, or concurrent renal impairment deemed unsuitable for serum albumin therapy by the investigator, such as diabetic kidney disease, hyperuricemia-related renal injury, sleep apnea-associated renal damage, hyperlipidemia-induced renal impairment, etc.;
5. Presence of severe underlying diseases at screening that the investigator deems inappropriate for study participation, including but not limited to active malignancy, pulmonary edema, bleeding tendencies or active bleeding disorders, uncontrolled infections (including spontaneous bacterial peritonitis), thyroid dysfunction (Grade 3 or higher according to the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE], version 5.0), etc.;
6. Positive for hepatitis B surface antigen (HBsAg), positive for hepatitis B core antibody (HBcAb) with detectable hepatitis B virus deoxyribonucleic acid (HBV-DNA), positive for hepatitis C antibody (HCV Ab) with detectable hepatitis C ribonucleic acid (HCV-RNA), positive for human immunodeficiency virus antibody (HIV Ab), or positive for Treponema pallidum (syphilis) antibodies at screening;
7. Presence of the following laboratory abnormalities at screening:

   * Liver function: Alanine transaminase (ALT) >3 times the upper limit of normal (ULN); Aspartate transaminase (AST) >3 ULN; Total bilirubin (TBIL) >1.5 ULN or deemed unsuitable for the trial by the investigator;
   * Renal function: Creatinine clearance (Ccr) <50 mL/min (calculated using the Cockcroft-Gault formula: Ccr(mL/min) = [(140 - age) × weight(kg)] / [72 × Scr(mg/dL)], multiplied by 0.85 for females);
   * Bone marrow function: Absolute neutrophil count (ANC) <1.5 × 10^9/L; Platelets (PLT) <100 × 10^9/L; Hemoglobin (HGB) <90 g/L;
8. History or presence of neurological disorders at screening, such as stroke, neuromyelitis optica, Parkinson's disease, epilepsy, etc.;
9. Patients with comorbid psychiatric disorders, including schizophrenia or other mental illnesses, bipolar disorder, depression, or delirium;
10. Contraindications to MRI scanning, including incompatible cardiac pacemakers/defibrillators, magnetic metal implants, etc.;
11. Irreversible visual or auditory impairments preventing completion of assessments related to cognition, neuropsychiatric symptoms, and activities of daily living;
12. Alcohol or drug abusers;
13. Pregnant or lactating women;
14. Received plasma derivatives (including human albumin) within 3 months prior to screening, history of organ transplantation, or planned to undergo invasive procedures or treatments during the study;
15. Participated in another clinical trial (excluding non-drug intervention trials) within 30 days prior to the screening visit for this trial or planning to participate in another trial during this study;
16. The investigator judges that the AD patient is unlikely to complete the trial, such as poor adherence to medication or scheduled visits.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The change in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) score from baseline to Week 25 post-treatment. | from baseline to Week 25 post-treatment

SECONDARY OUTCOMES:
The changes in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) scores from baseline at Weeks 7, 16, 29 (if applicable), 37 (if applicable), and 41 (if applicable) post-treatment. | At Weeks 7, 16, 25, 29 (if applicable), 37 (if applicable), and 41 (if applicable)
  The Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) is an instrument used to assess cognitive function in individuals with Alzheimer's disease or other forms of dementia. The scale ranges from 0 to 70, with lower scores indicating better cognitive function and higher scores indicating more severe cognitive impairment. Therefore, the lower the score on the ADAS-Cog, the better the cognitive performance of the individual being assessed. Conversely, a higher score indicates greater cognitive decline. The minimum possible score on the ADAS-Cog is 0, and the maximum possible score is 70.
The changes in Clinical Dementia Rating Scale - Global Score (CDR-GS) from baseline at Weeks 7, 16, 25, 29 (if applicable), 37 (if applicable), and 41 (if applicable) following treatment initiation. | At Weeks 7, 16, 25, 29 (if applicable), 37 (if applicable), and 41 (if applicable)
  The Clinical Dementia Rating - Global Score (CDR-GS) is a tool used by healthcare professionals to assess the severity of dementia in patients. The CDR-GS has a range from 0 to 3, with 0 representing no dementia, 0.5 indicating very mild dementia, 1 indicating mild dementia, 2 indicating moderate dementia, and 3 indicating severe dementia.
  Therefore, the lower the score on the CDR-GS, the better the cognitive and functional abilities of the individual being assessed. Conversely, a higher score indicates more severe dementia. The minimum possible score on the CDR-GS is 0, and the maximum possible score is 3.
The changes in Neuropsychiatric Inventory (NPI) scores from baseline at Weeks 7, 16, 25, 29 (if applicable), 37 (if applicable), and 41 (if applicable) after the commencement of treatment. | At Weeks 7, 16, 25, 29 (if applicable), 37 (if applicable), and 41 (if applicable)
  The Neuropsychiatric Inventory (NPI) is a tool used to evaluate neuropsychiatric symptoms in individuals with dementia. A lower score on the NPI indicates fewer or less severe neuropsychiatric symptoms, while a higher score suggests more frequent or severe symptoms. Thus, a lower NPI score is generally considered to be a better outcome. The minimum possible score is 0, and the maximum possible score is 144.
The changes in Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) ability assessment scale scores from baseline | At Weeks 7, 16, 25, 29 (if applicable), 37 (if applicable), and 41 (if applicable)
  The Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory (ADCS-ADL) is a tool designed to measure the functional ability of individuals with Alzheimer's disease. The ADCS-ADL has a range from 0 to 78, where 0 indicates complete dependence and 78 indicates complete independence. Higher scores on the ADCS-ADL indicate better functional status and ability to perform daily activities independently.ng the start of treatment.

OTHER OUTCOMES:
blood albumin concentration | At baseline (D0), 12 hours after the 5th dosing (W13D1), and 12 hours after the 9th dosing (W25D1)、12 hours following CSF collection
  Blood samples were collected and the concentration and quality of albumin in the blood were measured at baseline (D0), 12 hours after the 5th dosing (W13D1), and 12 hours after the 9th dosing (W25D1). Cerebrospinal Fluid (CSF) samples were collected during the treatment period (if CSF samples were obtained from the participants 12 hours after drug administration on W13D1 or W25D1, there was no need for repeated blood sampling).
oxidation level of serum albumin | At baseline (D0), 12 hours after the 5th dosing (W13D1), and 12 hours after the 9th dosing (W25D1)、12 hours following CSF collection
  including levels of free thiols, sulfonated residues, carbonylation, glycation, and homocysteinylation，These metrics will be compared against those of albumin from healthy individuals, ultimately deriving a paramete
cerebrospinal fluid albumin concentration | At baseline (D0) and 12 hours following any dosing event between W13D1 and W25D1 during the treatment period
  In each dose group, CSF (Cerebrospinal Fluid) samples are collected from at least 50% of the participants. The collection times are at baseline (D0) and 12 hours following any dosing event between W13D1 and W25D1 during the treatment period.
oxidation level of cerebrospinal fluid (CSF) albumin | At baseline (D0) and 12 hours following any dosing event between W13D1 and W25D1 during the treatment period
  including levels of free thiols, sulfonated residues, carbonylation, glycation, and homocysteinylation，These metrics will be compared against those of albumin from healthy individuals, ultimately deriving a paramete

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shang’ai, China

IPD SHARING:
Plan to Share IPD: No